CLINICAL TRIAL: NCT06671197
Title: Multicenter Randomized Controlled Study on Efficacy and Safety of Pulmonary Vein Isolation,Left Atrial Posterior Wall Ablation and Superior Vena Cava Isolation Using Pulsed Field Ablation for Persistent Atrial Fibrillation
Brief Title: Study on the Ablation of Persistent Atrial Fibrillation Using Pulsed Electric Fields Under Different Surgical Procedures
Status: Not yet recruiting | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 20240926
Record Dates: First submitted 2024-09-27; First posted 2024-11-04 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Persistent Atrial Fibrillation
Keywords: Pulsed Field Ablation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- PVI-only
  Interventions: Device: Pulmonary vein isolation
- PVI + PWI + SVCI: posterior left atrial wall isolation and superior vena cava isolation
  Interventions: Device: Pulmonary vein isolation+posterior left atrial wall line+superior vena cava isolation

INTERVENTIONS:
Device: Pulmonary vein isolation — Pulsed field ablation
  Groups: PVI-only
Device: Pulmonary vein isolation+posterior left atrial wall line+superior vena cava isolation — Pulsed field ablation
  Groups: PVI + PWI + SVCI

SUMMARY:
Atrial fibrillation (AF) is one of the most common arrhythmias in clinical practice, and there are more than 20 million AF patients in my country. Currently, rhythm control has become the main treatment option for AF, but there is still controversy over the best ablation procedure, especially whether other auxiliary ablation lines need to be added. Based on the existing clinical evidence, the durability and permeability of ablation damage are the main reasons for the differences. Pulsed electric field is a new ablation energy source based on the principle of cell electroporation. It has the characteristics of damage safety and permeability, so it is expected to solve the above dilemma. The study was divided into PVI (PVI-only) group according to the ratio of 1: 1, PVI + PWI + SVCI (posterior left atrial wall isolation and superior vena cava isolation) group. Through one-year follow-up of two groups of patients, the role of left atrial posterior wall and superior vena cava in the maintenance mechanism of persistent atrial fibrillation was explored, and the safety and effectiveness of domestic pulse ablation system were verified, which provided intellectual support for further medical and engineering integration

ELIGIBILITY:
Inclusion Criteria:

* 18 years old and above, regardless of gender;
* Patients with symptomatic drug-refractory persistent atrial fibrillation (diagnosis time exceeding ≤ 3 years);
* Agree to participate in the study and be able and willing to comply with all follow-up requirements;-

Exclusion Criteria:

* Left ventricular ejection fraction (LVEF) ≤ 35%
* Left atrial diameter (echocardiography) ≥ 55mm
* Patients with a definite thrombus in the left atrium or a definite thrombus in the heart before surgery
* Patients with cardiac function classification (NYHA) III-IV
* Patients with second-degree (type II) or third-degree atrioventricular block
* Persons with obvious congenital heart defects (such as atrial septal defect or severe pulmonary vein stenosis, but excluding patent foramen ovale)
* Patients with prosthetic valve implantation
* Patients with implanted cardiac pacemaker or cardiac defibrillator (ICD)
* Diagnosed with hypertrophic cardiomyopathy, chronic obstructive pulmonary disease, myxoma
* Patients with preoperatively known symptomatic carotid stenosis
* Patients with untreated or controlled hyperthyroidism or hypothyroidism
* Patients with systemically active infections
* Patients with renal failure who have significant bleeding tendency or are undergoing hemodialysis
* Patients with myocardial infarction or any cardiac intervention/open surgery within 3 months
* Patients who have had a stroke or transient ischemic attack within 6 months
* Patients with obvious contraindications to interventional surgery and who are judged by the investigator to be unable to undergo ablation surgery
* Women who are pregnant or breastfeeding or who have a family planning during the study period
* Patients who have participated in clinical trials of other drugs or medical devices within 3 months
* Patients considered inappropriate by the investigator to participate in this clinical trial -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1.18 years old and above, regardless of gender; 2.Patients with symptomatic drug-refractory persistent atrial fibrillation (diagnosis time exceeding ≤ 3 years); 3.Agree to participate in the study and be able and willing to comply with all follow-up requirements
Sampling Method: Probability Sample
Enrollment: 436 (Estimated)
Dates: Start 2025-03-31 (Estimated); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Surgical success rate | 12 months after surgery.
  Surgical success rate: Except for the blank period, there was no recurrence of atrial arrhythmia ≥30s within 12 months after surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Sichuan Jinjiang Electronic Medical Device Technology Co., Ltd, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Undecided
Undecided